CLINICAL TRIAL: NCT04633486
Title: Endoscopically One-year Follow-up in Patients After Small-bowel Transplantation, Role of SASAKI Score
Brief Title: Endoscopically One-year Follow-up in Patients After Small-bowel Transplantation
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 829/2020BO2
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Intestinal Graft Dysfunction
Keywords: endoscopic monitoring, intestinal transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: zoom-endoscopy — Endoscopic monitoring of intestinal transplant recipients is done with zoom-endoscopes for exact diagnostic of intestinal mucosa.
  Other Names: ZVE

SUMMARY:
Intestinal transplantation is associated with high numbers of ejection events. A close endoscopic controll of the intestinal graft is possible. Sasaki et al. presented 2002 an endoscopic score using zoom-endoscopes for early detection of rejection events.

DETAILED DESCRIPTION:
Small bowel transplantation is a potentially life-saving procedure for patients with irreversible gut failure, especially for those with total parenteral nutrition complications, inability to adapt to quality-of-life limitations posed by intestinal failure, and high risk of death if the native gut is not removed. Endoscopy provides the quickest method for assessing the overall health of graft mucosa and is essential in obtaining specimens from large areas for histologic evaluation, which continues to remain the gold standard for a diagnosis of rejection. Recently, the use of zoom videoendoscopy has been reported as a better evaluation of intestinal mucosa than the use of a standard endoscope. Acute cellular rejection in short-term follow-up, appears with acute and dramatic clinical symptoms (fever, vomiting, nausea, increased stomal output/diarrhea, abdominal pain, and distension), so that it is rarely predictable with surveillance.

Comparison of endoscopic and histo-pathologic findings should be performed.

ELIGIBILITY:
Inclusion Criteria:

* intestinal transplant recipients

Exclusion Criteria:

* younger age (< 16)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intestinal transplant reciepients since 2005
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Rate of congruent findings of zoom-endoscopy and pathological examinations | 12 months
  Reliability of zoom-endoscopy and pathological examinations

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided